CLINICAL TRIAL: NCT04946409
Title: Identification of Longitudinal Burden of Disease and Functional Impairment in X-Linked Hypophosphatemia
Brief Title: Burden of Disease and Functional Impairment in XLH
Acronym: IdeFIX
Status: Active, not recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IdeFIX
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: X Linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum / Plasma / Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Observational study comprising prospective follow up as well as retrospective chart review in order to evaluate the longitudinal course of the disease in XLH patients with a specific focus on functional impairment, physical performance and complications associated with the disease or respective treatment.

DETAILED DESCRIPTION:
This is an observational / non-interventional study in order to assess the longitudinal course of XLH including disease related burden of disease and functional impairment. This is accomplished by both prospective follow up of affected patients as well as retrospective chart review. Evaluation conducted as per clincal routine and specifically evaluated as part of this study will include

* baseline documententation / demographic (as obtained from medical records)
* general data on XLH-disease specific medical history
* physical examination results
* functional assessments
* technical assessments
* quality of life / questionnaires
* laboratory evaluations

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years, inclusive, at the time of enrollment
* Diagnosis of X-linked Hypophosphatemia confirmed by

  * documented PHEX mutation in either the patient, or in a directly related family member
  * positive family history of XLH and symptoms of the disease or
  * Phosphaturia + elevated serum levels of c-term FGF23 or iFGF23 and symptoms of the disease
* Written informed consent

Exclusion Criteria:

- Suspected of confirmed diagnosis of another phosphate wasting disorder

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with X-linked Hypophosphatemia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Course of disease | retrospective and up to 48 months from enrollment
  To document and assess the natural course of disease, associated symptoms and functional impairment in adult patients with XLH.

SECONDARY OUTCOMES:
Comorbidities and medical treatment | retrospective and up to 48 months from enrollment
  Assess and document comorbidities and medical treatment regimens applied in adult patients with XLH
Functional deficits and mobility constraints | retrospective and up to 48 months from enrollment
  Assess and document functional deficits and mobility constraints in adult patients with XLH
Laboratory values | retrospective and up to 48 months from enrollment
  Assess laboratory parameters over time in adults with XLH
Organ / tissue specific health issues | retrospective and up to 48 months from enrollment
  Describe frequency and outcome of organ / tissue specific health issues (affecting e.g. skeleton, dental health, muscles and joints) in adults with XLH
Safety and tolerability of treatment | retrospective and up to 48 months from enrollment
  Evaluate safety and tolerability of various treatment regimens commonly applied in XLH patients
Quality of life | retrospective and up to 48 months from enrollment
  Assess quality of life and respective determining factors in adults patients with XLH

OTHER OUTCOMES:
Impact of treatment on physical performance | retrospective and up to 48 months from enrollment
  Evaluate the impact of clinical routine treatment including both medical approaches and physical therapy on physical performance and mobility of adult patients with XLH
Medical history | retrospective and up to 48 months from enrollment
  Document and assess medical history of adult patients with XLH in order to understand its predictive value on burden of disease in adulthood

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Center for Musculoskeletal Research, Orthopedic Department, University of Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared in order to warrant patients privacy.